CLINICAL TRIAL: NCT01430845
Title: Predicting Developmental Disability Type and Mental Retardation Level in Children Who Were Diagnosed in General Developmental Delay
Brief Title: Predicting Developmental Disability Type and Mental Retardation Level in Children With General Developmental Delay
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: SHEBA-11-8458-LG-CTIL
Record Dates: First submitted 2011-09-07; First posted 2011-09-08 (Estimated); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Global Developmental Delay; Cerebral Palsy; Mental Retardation; Pervasive Developmental Disorders
Keywords: GDD; CP; MR; PDD; ASD; BSID
MeSH Terms: conditions — Learning Disabilities; Cerebral Palsy; Intellectual Disability; Child Development Disorders, Pervasive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to find the relationship between the stage and quality of developmental delay during infancy and toddler age, and the final diagnosis that the child gets a few years later (MR, type of PDD, CP or comorbidity of a few disorders).

DETAILED DESCRIPTION:
The purpose of this study is to find the relationship between the stage and quality of developmental delay at a young age, and the final diagnosis that the child gets a few years later (MR, type of PDD, CP or comorbidity of a few disorders). We assume that analysis of developmental subtests can show the developmental direction of the child and predict his later diagnosis. The developmental test which is chosen for this purpose is the BSID which is a comprehensive and worldwide developmental test. In addition, we want to find the correlation between the developmental delays in early age and the intellectual functioning in the future. We assume that through analyzing the subtests of developmental tests we will succeed in predicting the expected cognitive level (IQ).

Medical files of participating children will be analyzed. The files will be sorted and only those of GDD diagnosis containing BSID test data will be selected. The performances of the BSID test and the current diagnosis of the children will be recorded. A trained researcher will process the BSID data and build a database which will include the findings of the test, the current diagnosis of the child and the level of MR, in case the child suffers from MR (only or comorbidly). In order to test the research assumptions appropriate statistic tests will be done using the statistical program SPSS version 17.

This study has important implications. Findings which show that the developmental tests are effective tools, not only to evaluate general developmental delay, but as auxiliary tools for diagnosing and predicting the type of disability and level of retardation. These findings are a breakthrough in the diagnostic field. In addition, the ability to predict the type of disability and level of mental retardation by a developmental test that is used so widely allows early intervention, and as has been widely proven, the earlier the intervention, the better the outcome.

In addition, a vast range of people will benefit from the findings. Professionals such as doctors, psychologists and paramedical therapists, government bodies and community resources that can design and build a support system and services for the child and his family. Most importantly, the family of the diagnosed child and the child himself will be able to prepare themselves to the new reality and design their life accordingly.

ELIGIBILITY:
Inclusion Criteria:

* GDD diagnosis in two axis' at least
* BSID test in its second or third version

Exclusion Criteria:

* If not all of the data is available for all of the assessments

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will be conducted at the Child Development Center in Tel-Hashomer hospital (Ramat-Gan, Israel). The target population is all children who were diagnosed at the hospital with GDD (in two axis' at least) between the years 2003 to 2005. They must also have undergone the BSID test in its second or third version. The data must be available on all assessments (N~150). The children were 1.5-3 years old at diagnosis and diagnosed by a doctor and psychologist. Today these children are 5-7 years old. Some of them are still being treated in Tel-Hashomer. The children live all over the country
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2011-09-01; Primary Completion 2015-12-01 (Actual); Study Completion 2015-12-01 (Actual)

PRIMARY OUTCOMES:
level of Mental retardation in older age | non

CONTACTS AND LOCATIONS:
Overall Officials: Lidia Gabis, MD, Principal Investigator — Sheba Medical Center; Shefer Shahar, PHD, Study Director — Sheba Medical Center; Bat Chen Amir, BA, Study Director — Sheba Medical Center
Locations (1):
- Weinberg Child Development Center, Sheba Medical Center, Tel-Hashomer, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Undecided